CLINICAL TRIAL: NCT06249243
Title: Patterns of Renal & Urinary Involvement in Patients With Inflammatory Bowel Diseases Who Attended to Assiut University Hospitals
Brief Title: Affection of Renal and Urinary System in IBD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rania Essam Mohamed, Assistant Lecturer, Assiut University
Other Study IDs: Renal and urinary in IBD
Record Dates: First submitted 2023-12-09; First posted 2024-02-08 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Nephrolithiasis, Glomerulonephritis, Amyloidosis,AKI, CKD, Tubuli Interstitial; Urinary System Disorders in IBD Patients
MeSH Terms: conditions — Nephrolithiasis; Glomerulonephritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Detection and classification of different renal and urinary affection in patients with IBD that attended to Assist University Hospitals

DETAILED DESCRIPTION:
Background (Research Question, Available Data from the literature, Current strategy for dealing with the problem, Rationale of the research that paves the way to the aim(s) of the work). (200-250 words max.) Inflammatory bowel disease is an idiopathic disease cause sever inflammation of GIT , presentes in ulcerative colitis or Crohn's disease occur in 6%-47%

IBD is profoundly associated with extra intestinal manifestions , Especially renal and urinary involvement occurs in 4% - 23% of patients with IBD.

Patterns of renal complications include nephrolithiasis, glomerulonephritis, amyloidosis, AKl, CKD, tubulointerstitial nephritis, asymptomatic proteinuria and hematuria; each type has specific mechanism

Nephrolithiasis is 10-100 times greater in IBD patients than general population.most common stones are calcium, oxalate and urate; Stones occur due to loss of electrolytes "Mg,k" due to diarrhea which lead to crystallization.

Glomerulonephritis pattern in IBD , is associated with IgA nephropathy, IgM nephropathy, membranous and focal segmental glomerulonephritis.

There is genetic connection between IgA nephropathy and intestinal diseases!

Secondary amyloidosis (AA-type) is a rare but serious complication of IBD.renal amyloidosis had been proven to be the most common lethal manifestion of IBD - associated amyloidosis (A), since renal involvement rapidly leads to end stage renal failure.

Sever long -standing IBD consists a predisposing factor for renal complications that occur in 4-23 % of patients So we aim to shed more light on the pathophysiology of renal damage in IBD; considering the renal manifestions and complications of IBD, it is important to emphasize the role of screening of renal function in preventing, diagnosing, and,if possible, reversing probable kidney damage.

ELIGIBILITY:
Inclusion Criteria:

* 100 patients suffering of IBD who attended to AUH either with Crohn's or ulcerative colitis with different presentation

Exclusion Criteria:

* Patients with other known cause of kidney or urinary affection as DM,HTN,APCKD, lupus nephritis,UTI…..

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Sample size was calculated by using it open -epi version 3 According to the prevalence of urinary affection in IBD patients 13,5%() Sample size was 92 patient at confidance level 95% +-7 confidance limit
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
Patterns of renal and urinary involvement in IBD patients | 2 years
  Is renal and urinary system affect on IBD patients ?